CLINICAL TRIAL: NCT05859555
Title: Multimodal Educative Data Feedback for Deprescribing Benzodiazepine (BZD) and Related Drugs in Outpatients: a Cluster Randomized Controlled Study
Brief Title: Multimodal Educative Data Feedback for Deprescribing BZD and Related Drugs in Outpatients: a Cluster RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Réseau de soins Delta (Other)
Responsible Party: Principal Investigator, Minette-Joëlle Zeukeng, Project Manager, Réseau de soins Delta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BZD001
Record Dates: First submitted 2023-03-19; First posted 2023-05-16 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Deprescription; Benzodiazepine (BZD) and Related Drugs
Keywords: Benzodiazepine (BZD) and related drugs; Deprescribing; Safety; Older patients

STUDY DESIGN:
Intervention Model Description: Cluster randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Thematic quality circles - Deprescription (Other)
  Interventions: Other: Thematic quality circles - Deprescription
- No intervention (No Intervention)

INTERVENTIONS:
Other: Thematic quality circles - Deprescription — Thematic quality circles on benzodiazepines and analogues with a pharmacist (practical cases)
  Arms: Intervention: Thematic quality circles - Deprescription

SUMMARY:
Benzodiazepine (BZD) and related drugs are sedative anxiolytics and hypnotics that should be avoided especially in people aged 65 years and older, given the high risk of falling, fracture, dependence, respiratory depression and cognitive disorders. Despite these contraindications, their consumption continues to increase in Switzerland.

Although it can be assumed that deprescribing a drug has a direct benefit, it is nevertheless necessary to determine how to implement this process effectively and safely. To change healthcare professionals' prescribing behaviours for BZD, the most common deprescribing interventions include identification of appropriate patients, education and training of GPs and patients, and gradual and appropriate reduction of the dose of BZD. Thus, the DELTA CARE NETWORK and the DELTA VAUD CARE NETWORK have set themselves the task of evaluating the effectiveness of a multimodal deprescribing intervention for Delta primary care physicians and their patients aged 65 and over, in the cantons of Geneva and Vaud. The goal is to reduce the total BZD prescription rate among this population.

This quality development project is fully in line with the Quality Federal Commission's objectives of efficiency, safety, patient-centred and in the interests of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Physician who attended a quality cercle in the cantons of Geneva and Vaud
* Prescribed at least one prescription of Benzodiazepines during the year of analysis to patient aged 65 years and older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Rate Benzodiazepine (BZD) and related drugs prescribed by primary care physicians | 9 months
  Reduce the total BZD prescribing frequency by 20% 9 months after the interventioncompared to the control group (DDD/1000 patients over 9 months). The drug measure will be the DDD daily dose defined by the World Health Organization Collaborating Centre for Drug Statistics Methodology (or number of tablets or number of packages).

SECONDARY OUTCOMES:
Rate of patients aged 65 years who took long-term BZD | 18 months
  Reduce by 20% the prevalence of 65-year-old patients with long-term use (more than 3 months) of BZD as well as the prevalence of long-term users 18 months after intervention (number of BDZ patients per physician/QC per year).

CONTACTS AND LOCATIONS:
Locations (1):
- Réseau de soins Delta SA, Geneva, Petit Lancy, Switzerland

IPD SHARING:
Plan to Share IPD: No